CLINICAL TRIAL: NCT03877081
Title: Effect of Probiotics and Prebiotics in Renal Function in Septic Acute Kidney Injury Patients, Randomized Control Trial
Brief Title: Effect of Probiotics and Prebiotics in Renal Function in Septic Acute Kidney Injury Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Jonathan Samuel Chavez Iñiguez, MD, Nephrologist, Principal investigator, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AKI and Probiotics
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Acute Kidney Injury; Probiotics; Sepsis
Keywords: Acute kidney injury; Probiotics; Sepsis; Shock
MeSH Terms: conditions — Acute Kidney Injury; Sepsis; Shock | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotics. Intervention patients (Experimental): This patients will receive 2 doses of oral probiotics a day, for seven days
  Interventions: Biological: Probiotics
- Placebo group (Placebo Comparator): This patients will receive 2 doses of oral placebo a day, for seven days
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Probiotics — Administration of oral probiotics with 2 doses a day
  Arms: Probiotics. Intervention patients
Other: Placebo — Administration of oral placebo with 2 doses a day
  Arms: Placebo group

SUMMARY:
Septic acute kidney injury is a condition associated with highly related to inflammatory molecules. Prebiotics and probiotics have shown to improve inflammatory cascade in animal model; In this study, the investigators propose the use of probiotics to improve the clinical evolution of septic acute kidney injury patients.

DETAILED DESCRIPTION:
Acute kidney injury is most commonly caused by sepsis, where endotoxemia and an expanding inflammatory reaction play a key role in its pathogenesis, when this condition is present it is highly related to poor clinical outcomes and higher mortality rates. There is no current specific treatment, and the therapeutic approach is more orientated to complication management. In this study, the investigators propose the use of probiotics to improve the clinical evolution of septic acute kidney injury patients.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis by SOFA
* Acute kidney injury by KDIGO

Exclusion Criteria:

* No presence of sepsis
* No presence of AKI
* Age below 18 years
* Inability or contraindication for oral capsules or probiotics by nasogastric tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2022-09-04 (Estimated); Study Completion 2023-02-04 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine | 7 days
  Number of participants with significative reduction of serum creatinine concentration from beginning of the intervention

SECONDARY OUTCOMES:
Death | 7 days
  Number of defunctions among the subjects
Renal replacement therapy | 7 days
  Number of participants that initiate renal replacement therapy
Final creatinine | 7 days
  Last recorded serum creatinine concentration
Urinary output (final) | 7 days
  Quantification of urinary output in ml/Kg/hour
Shock days | 7 days
  Use of vasopressor therapy during hospitalization
Recuperation of basal creatinine | 7 days
  Serum creatinine reduction to 25% from basal creatinine
Length of hospitalization | 7 days
  Days of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- HCG, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lameire NH, Bagga A, Cruz D, De Maeseneer J, Endre Z, Kellum JA, Liu KD, Mehta RL, Pannu N, Van Biesen W, Vanholder R. Acute kidney injury: an increasing global concern. Lancet. 2013 Jul 13;382(9887):170-9. doi: 10.1016/S0140-6736(13)60647-9. Epub 2013 May 31. PMID 23727171
- [Background] Siew ED, Davenport A. The growth of acute kidney injury: a rising tide or just closer attention to detail? Kidney Int. 2015 Jan;87(1):46-61. doi: 10.1038/ki.2014.293. Epub 2014 Sep 17. PMID 25229340
- [Background] Murugan R, Karajala-Subramanyam V, Lee M, Yende S, Kong L, Carter M, Angus DC, Kellum JA; Genetic and Inflammatory Markers of Sepsis (GenIMS) Investigators. Acute kidney injury in non-severe pneumonia is associated with an increased immune response and lower survival. Kidney Int. 2010 Mar;77(6):527-35. doi: 10.1038/ki.2009.502. Epub 2009 Dec 23. PMID 20032961
- [Background] Nisula S, Kaukonen KM, Vaara ST, Korhonen AM, Poukkanen M, Karlsson S, Haapio M, Inkinen O, Parviainen I, Suojaranta-Ylinen R, Laurila JJ, Tenhunen J, Reinikainen M, Ala-Kokko T, Ruokonen E, Kuitunen A, Pettila V; FINNAKI Study Group. Incidence, risk factors and 90-day mortality of patients with acute kidney injury in Finnish intensive care units: the FINNAKI study. Intensive Care Med. 2013 Mar;39(3):420-8. doi: 10.1007/s00134-012-2796-5. Epub 2013 Jan 5. PMID 23291734
- [Background] Bagshaw SM, George C, Dinu I, Bellomo R. A multi-centre evaluation of the RIFLE criteria for early acute kidney injury in critically ill patients. Nephrol Dial Transplant. 2008 Apr;23(4):1203-10. doi: 10.1093/ndt/gfm744. Epub 2007 Oct 25. PMID 17962378
- [Background] Ostermann M, Chang RW. Acute kidney injury in the intensive care unit according to RIFLE. Crit Care Med. 2007 Aug;35(8):1837-43; quiz 1852. doi: 10.1097/01.CCM.0000277041.13090.0A. PMID 17581483
- [Background] Hoste EA, Clermont G, Kersten A, Venkataraman R, Angus DC, De Bacquer D, Kellum JA. RIFLE criteria for acute kidney injury are associated with hospital mortality in critically ill patients: a cohort analysis. Crit Care. 2006;10(3):R73. doi: 10.1186/cc4915. Epub 2006 May 12. PMID 16696865
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Background] Chawla LS, Amdur RL, Amodeo S, Kimmel PL, Palant CE. The severity of acute kidney injury predicts progression to chronic kidney disease. Kidney Int. 2011 Jun;79(12):1361-9. doi: 10.1038/ki.2011.42. Epub 2011 Mar 23. PMID 21430640
- [Background] Wang HE, Muntner P, Chertow GM, Warnock DG. Acute kidney injury and mortality in hospitalized patients. Am J Nephrol. 2012;35(4):349-55. doi: 10.1159/000337487. Epub 2012 Apr 2. PMID 22473149
- [Background] Zarjou A, Agarwal A. Sepsis and acute kidney injury. J Am Soc Nephrol. 2011 Jun;22(6):999-1006. doi: 10.1681/ASN.2010050484. Epub 2011 May 12. PMID 21566052
- [Background] Gomez H, Ince C, De Backer D, Pickkers P, Payen D, Hotchkiss J, Kellum JA. A unified theory of sepsis-induced acute kidney injury: inflammation, microcirculatory dysfunction, bioenergetics, and the tubular cell adaptation to injury. Shock. 2014 Jan;41(1):3-11. doi: 10.1097/SHK.0000000000000052. PMID 24346647
- [Background] Mehta RL, Bouchard J, Soroko SB, Ikizler TA, Paganini EP, Chertow GM, Himmelfarb J; Program to Improve Care in Acute Renal Disease (PICARD) Study Group. Sepsis as a cause and consequence of acute kidney injury: Program to Improve Care in Acute Renal Disease. Intensive Care Med. 2011 Feb;37(2):241-8. doi: 10.1007/s00134-010-2089-9. Epub 2010 Dec 9. PMID 21152901
- [Background] Peters E, Antonelli M, Wittebole X, Nanchal R, Francois B, Sakr Y, Vincent JL, Pickkers P. A worldwide multicentre evaluation of the influence of deterioration or improvement of acute kidney injury on clinical outcome in critically ill patients with and without sepsis at ICU admission: results from The Intensive Care Over Nations audit. Crit Care. 2018 Aug 3;22(1):188. doi: 10.1186/s13054-018-2112-z. PMID 30075798
- [Background] Bellomo R, Kellum JA, Ronco C, Wald R, Martensson J, Maiden M, Bagshaw SM, Glassford NJ, Lankadeva Y, Vaara ST, Schneider A. Acute kidney injury in sepsis. Intensive Care Med. 2017 Jun;43(6):816-828. doi: 10.1007/s00134-017-4755-7. Epub 2017 Mar 31. PMID 28364303
- [Background] Gomez H, Kellum JA. Sepsis-induced acute kidney injury. Curr Opin Crit Care. 2016 Dec;22(6):546-553. doi: 10.1097/MCC.0000000000000356. PMID 27661757
- [Background] Dellepiane S, Marengo M, Cantaluppi V. Detrimental cross-talk between sepsis and acute kidney injury: new pathogenic mechanisms, early biomarkers and targeted therapies. Crit Care. 2016 Mar 15;20:61. doi: 10.1186/s13054-016-1219-3. PMID 26976392
- [Background] Mariano F, Cantaluppi V, Stella M, Romanazzi GM, Assenzio B, Cairo M, Biancone L, Triolo G, Ranieri VM, Camussi G. Circulating plasma factors induce tubular and glomerular alterations in septic burns patients. Crit Care. 2008;12(2):R42. doi: 10.1186/cc6848. Epub 2008 Mar 25. PMID 18364044
- [Background] Pickkers P, Ostermann M, Joannidis M, Zarbock A, Hoste E, Bellomo R, Prowle J, Darmon M, Bonventre JV, Forni L, Bagshaw SM, Schetz M. The intensive care medicine agenda on acute kidney injury. Intensive Care Med. 2017 Sep;43(9):1198-1209. doi: 10.1007/s00134-017-4687-2. Epub 2017 Jan 30. PMID 28138736
- [Background] Cigarran Guldris S, Gonzalez Parra E, Cases Amenos A. Gut microbiota in chronic kidney disease. Nefrologia. 2017 Jan-Feb;37(1):9-19. doi: 10.1016/j.nefro.2016.05.008. Epub 2016 Aug 21. English, Spanish. PMID 27553986
- [Background] Vanholder R, Glorieux G. The intestine and the kidneys: a bad marriage can be hazardous. Clin Kidney J. 2015 Apr;8(2):168-79. doi: 10.1093/ckj/sfv004. Epub 2015 Feb 10. PMID 25815173
- [Background] Ranganathan N, Friedman EA, Tam P, Rao V, Ranganathan P, Dheer R. Probiotic dietary supplementation in patients with stage 3 and 4 chronic kidney disease: a 6-month pilot scale trial in Canada. Curr Med Res Opin. 2009 Aug;25(8):1919-30. doi: 10.1185/03007990903069249. PMID 19558344
- [Background] Icaza-Chavez ME. [Gut microbiota in health and disease]. Rev Gastroenterol Mex. 2013 Oct-Dec;78(4):240-8. doi: 10.1016/j.rgmx.2013.04.004. Epub 2013 Nov 28. Spanish. PMID 24290319
- [Background] Vaziri ND, Wong J, Pahl M, Piceno YM, Yuan J, DeSantis TZ, Ni Z, Nguyen TH, Andersen GL. Chronic kidney disease alters intestinal microbial flora. Kidney Int. 2013 Feb;83(2):308-15. doi: 10.1038/ki.2012.345. Epub 2012 Sep 19. PMID 22992469
- [Background] Natarajan R, Pechenyak B, Vyas U, Ranganathan P, Weinberg A, Liang P, Mallappallil MC, Norin AJ, Friedman EA, Saggi SJ. Randomized controlled trial of strain-specific probiotic formulation (Renadyl) in dialysis patients. Biomed Res Int. 2014;2014:568571. doi: 10.1155/2014/568571. Epub 2014 Jul 24. PMID 25147806
- [Background] Miranda Alatriste PV, Urbina Arronte R, Gomez Espinosa CO, Espinosa Cuevas Mde L. Effect of probiotics on human blood urea levels in patients with chronic renal failure. Nutr Hosp. 2014 Mar 1;29(3):582-90. doi: 10.3305/nh.2014.29.3.7179. PMID 24559003
- [Background] Koppe L, Mafra D, Fouque D. Probiotics and chronic kidney disease. Kidney Int. 2015 Nov;88(5):958-66. doi: 10.1038/ki.2015.255. Epub 2015 Sep 16. PMID 26376131
- [Background] Wanchai K, Pongchaidecha A, Chatsudthipong V, Chattipakorn SC, Chattipakorn N, Lungkaphin A. Role of Gastrointestinal Microbiota on Kidney Injury and the Obese Condition. Am J Med Sci. 2017 Jan;353(1):59-69. doi: 10.1016/j.amjms.2016.11.019. Epub 2016 Nov 17. PMID 28104104
- [Background] Yoshifuji A, Wakino S, Irie J, Tajima T, Hasegawa K, Kanda T, Tokuyama H, Hayashi K, Itoh H. Gut Lactobacillus protects against the progression of renal damage by modulating the gut environment in rats. Nephrol Dial Transplant. 2016 Mar;31(3):401-12. doi: 10.1093/ndt/gfv353. Epub 2015 Oct 20. PMID 26487672
- [Background] Taki K, Takayama F, Niwa T. Beneficial effects of Bifidobacteria in a gastroresistant seamless capsule on hyperhomocysteinemia in hemodialysis patients. J Ren Nutr. 2005 Jan;15(1):77-80. doi: 10.1053/j.jrn.2004.09.028. PMID 15648012
- [Background] Takayama F, Taki K, Niwa T. Bifidobacterium in gastro-resistant seamless capsule reduces serum levels of indoxyl sulfate in patients on hemodialysis. Am J Kidney Dis. 2003 Mar;41(3 Suppl 1):S142-5. doi: 10.1053/ajkd.2003.50104. PMID 12612972
- [Background] Ando Y, Miyata Y, Tanba K, Saito O, Muto S, Kurosu M, Homma S, Kusano E, Asano Y. [Effect of oral intake of an enteric capsule preparation containing Bifidobacterium longum on the progression of chronic renal failure]. Nihon Jinzo Gakkai Shi. 2003;45(8):759-64. Japanese. PMID 14737993
- [Background] Ogawa T, Shimada M, Nagano N, Ito K, Ando T, Shimomura Y, Ando Y, Otsuka K. Oral administration of Bifidobacterium longum in a gastro-resistant seamless capsule decreases serum phosphate levels in patients receiving haemodialysis. Clin Kidney J. 2012 Aug;5(4):373-4. doi: 10.1093/ckj/sfs072. No abstract available. PMID 25874106
- [Background] Yang J, Summanen PH, Henning SM, Hsu M, Lam H, Huang J, Tseng CH, Dowd SE, Finegold SM, Heber D, Li Z. Xylooligosaccharide supplementation alters gut bacteria in both healthy and prediabetic adults: a pilot study. Front Physiol. 2015 Aug 7;6:216. doi: 10.3389/fphys.2015.00216. eCollection 2015. PMID 26300782
- [Background] Finegold SM, Li Z, Summanen PH, Downes J, Thames G, Corbett K, Dowd S, Krak M, Heber D. Xylooligosaccharide increases bifidobacteria but not lactobacilli in human gut microbiota. Food Funct. 2014 Mar;5(3):436-45. doi: 10.1039/c3fo60348b. PMID 24513849
- [Background] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Derived] Chavez-Iniguez JS, Ibarra-Estrada M, Gallardo-Gonzalez AM, Cisneros-Hernandez A, Claure-Del Granado R, Chavez-Alonso G, Hernandez-Barajas EM, Romero-Munoz AC, Ramos-Avellaneda F, Prieto-Magallanes ML, Plascencia-Cruz M, Tanaka-Gutierrez JA, Perez-Hernandez C, Navarro-Blackaller G, Medina-Gonzalez R, Alcantar-Vallin L, Renoirte-Lopez K, Garcia-Garcia G. Probiotics in septic acute kidney injury, a double blind, randomized control trial. Ren Fail. 2023;45(2):2260003. doi: 10.1080/0886022X.2023.2260003. Epub 2023 Sep 19. PMID 37724527